CLINICAL TRIAL: NCT06373848
Title: The Impact of Vitamin E and CoQ10 Supplements as an Adjunctive Non-surgical Periodontal Therapy on Chronic Periodontitis and Salivary Markers.
Brief Title: Non-surgical Treatment of Chronic Periodontitis With an Adjunctive Vitamin E and Coenzyme Q10 Supplementation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Islamic Azad University, Sanandaj (Other)
Responsible Party: Principal Investigator, Amirhossein Farahmand, Periodontist, Associate Professor, Department of Periodontics, Faculty of Dentistry, Tehran Medical Sciences, Islamic Azad University, Tehran, Iran, Affiliation: Islamic Azad University, Tehran, Islamic Azad University, Sanandaj
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 346
Record Dates: First submitted 2024-04-16; First posted 2024-04-18 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Periodontal Diseases
Keywords: Periodontal disease, CoQ10, Vitamin E, antioxidant, saliva.
MeSH Terms: conditions — Periodontal Diseases | interventions — coenzyme Q10; Vitamin E

STUDY DESIGN:
Intervention Model Description: Parallel Assignment, Randomized, Double-blind, Controlled design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study was carried out utilizing a double-blind approach. In order to guarantee objectivity, all three groups - the Vitamin E group, the Coq10 group, and the control group - received medications that were indistinguishable in terms of appearance, packaging, and color. Additionally, to minimize any potential bias, a clinician who had no association with the research labeled the medications as A, B, and C (empty) based on their content, and then distributed them among the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vitamin E (Experimental): Participants in Group A were administered 400 mg of Vitamin E supplements on a daily basis throughout the two-month study period. After the study concluded, the clinical periodontal parameters were reevaluated to assess any potential impact of the supplements on oral health.. To compare the total antioxidant capacity in saliva before and after the consumption of the Vitamin E supplements, as well as in individuals who did not receive any form of medication, 2 ml of non-stimulated saliva was collected from each participant at the commencement and conclusion of the study. These samples were then analyzed using UV-spectrophotometric methods to determine any variations in antioxidant levels.
  Interventions: Drug: Receive 30 mg of Coq10
- Coq10 (Experimental): Participants in Group B were administered a daily dose of 30 mg of Coq10 supplements for two months. Following the study period, the clinical periodontal parameters were reevaluated to assess any potential impact of the supplements on oral health. To compare the total antioxidant capacity of saliva before and after the consumption of Coq10 supplements, as well as in individuals who did not receive any medication, 2 ml of non-stimulated saliva was collected from each participant at the commencement and conclusion of the study. The collected samples were then analyzed using UV-spectrophotometric methods to determine any variations in antioxidant levels.
  Interventions: Drug: Receive 30 mg of Coq10
- no-medication; (Active Comparator): Group C was not administered any medication during the study period lasting two months. Following this period, the clinical periodontal parameters were evaluated once again. Moreover, to analyze the total antioxidant capacity in saliva before and after the consumption of these supplements, as well as in individuals who were not given any medication, 2 ml of non-stimulated saliva was gathered from every participant at the commencement and conclusion of the study. This analysis was conducted using UV-spectrophotometric techniques.
  Interventions: Drug: Receive 30 mg of Coq10

INTERVENTIONS:
Drug: Receive 30 mg of Coq10 — A total of 120 individuals diagnosed with chronic periodontitis were selected for this study. These participants were randomly assigned to two different groups. The purpose of the study was to measure the periodontal parameters of the two molars adjacent to the mandible using a periodontal probe. All of the patients received scaling and root planing (SRP) as part of their treatment. However, the treatment groups differed in terms of the supplements they received. Group A was given a daily dose of Coq10 at 30 mg, while Group B received a daily dose of Vitamin E at 400 mg; Furthermore, group C did not receive any supplements. The periodontal examination involved a total of 300 teeth across the three groups. In addition to this, 2 ml of unstimulated saliva was collected from each patient both before and after 2 months. The purpose of collecting the saliva samples was to evaluate the total antioxidant capacity and determine if there were any changes over time.
  Other Names: Receive 400 mg of Vitamin E; non Receive any medication

SUMMARY:
Non-surgical treatment of chronic periodontitis with vitamin E and coenzyme Q10 supplementation

DETAILED DESCRIPTION:
This research was structured as a double-blind, randomized clinical trial to assess the effectiveness of CoQ10 and Vitamin E supplements on periodontal health in patients with chronic periodontitis. A total of 120 patients from the Department of Periodontics at Boroujerd Dental School of the Islamic Azad University of Medical Sciences were chosen for the study. Before the commencement of the trial, various clinical periodontal parameters such as plaque index, bleeding on probing, gingival index, probing depth, and clinical attachment level were measured in six different areas of the tooth surface. Subsequently, scaling and root planning were carried out, and oral hygiene practices were enhanced for all participants. The participants were then randomly divided into three groups: Group A received 30 mg of CoQ10, Group B received 400 mg of Vitamin E supplements daily, and Group C did not receive any medication. After two months, the clinical periodontal parameters were reevaluated. Furthermore, to compare the total antioxidant capacity in saliva before and after the administration of these supplements, as well as in patients who did not receive any medication, 2 ml of non-stimulated saliva was collected from each participant at the beginning and end of the study for analysis using UV-spectrophotometric methods. The selection criteria for eligible participants in this study were also clearly defined.

ELIGIBILITY:
Inclusion Criteria:

healthy individuals, between the ages of 28 and 35, there is a presence of chronic initial periodontal disease, now categorized as Stage-I, with a maximum pocket depth of 5 mm, specifically affecting the mandibular molar teeth in every quadrant.

Exclusion Criteria:

Conditions that may affect orthodontic treatments include systemic diseases, ongoing orthodontic treatments, pregnancy and breastfeeding, and the use of medications that can impact the periodontium, such as antibiotics, within the past 6 months. Additionally, recent malignancy, radiotherapy, or chemotherapy within the past 5 years can also have an impact. It is important to consider factors such as plaque index and bleeding scores, which should be below 25%, as well as any history of periodontal surgery at the desired treatment site within the past 6 months. Furthermore, the use of medicinal supplements within the past 6 months and cigarette smoking or tobacco use should also be taken into account.

Eligibility Criteria:

The study population consisted of 80 eligible individuals who were enrolled in this research project, which was specifically designed to conduct Randomized Double-Blind Clinical Trials.

Ages: 28 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Total Antioxidant capacity (TAC) of saliva | 3 months
  UV-spectrophotometry was employed to assess the overall antioxidant capacity in saliva before and after the consumption of these supplements, as well as in individuals who were not administered any medication. A total of 2 ml of non-stimulated saliva was collected from each participant at the commencement and conclusion of the study for analysis using UV-spectrophotometric techniques. Additionally, the selection of eligible participants for dis study was determined based on the following criteria.

SECONDARY OUTCOMES:
Bleeding on probing | 3 months
  The evaluation of the bleeding index will involve the utilization of a periodontal probe, which will be used to compare the results with other groups at the beginning and end of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Amirhossein Farahmand, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes
find great satisfaction in the availability of individual participant data sets for sharing. These IPS serve as the foundation for published results and can be easily shared with others.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3 Months